CLINICAL TRIAL: NCT00423644
Title: A Phase II Trial of ZIO-101 in Advanced Multiple Myeloma: Protocol SGL2001b
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL2001b
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; arsenic; cancer study; failed treatment
MeSH Terms: conditions — Multiple Myeloma | interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Darinaparson

INTERVENTIONS:
Drug: Darinaparson — 420 mg/m2 of Darinaparsin given twice weekly for three weeks, followed by one week of rest for up to six months
  Other Names: ZIO-101

SUMMARY:
The study of safety of a new organic arsenic compound in the treatment of advanced multiple myeloma

ELIGIBILITY:
Inclusion Criteria

1. Subjects with a confirmed diagnosis of active multiple myeloma with measurable protein criteria present to evaluate response. Measurable disease is defined as having at least one of the following criteria within 28 days prior to registration:

   1. Serum M-protein level > 0.5 gm/dl (10.0 g/L) measured by serum protein electrophoresis.
   2. Urinary M-protein excretion > 0.2 g/24 hours by urine electrophoresis.
2. Subjects must have relapsed or resistant disease, defined as either relapsing or is resistant after > 2 lines of prior therapy for myeloma. A minimum of 42 days must have elapsed since prior autologous or allogeneic transplant;
3. Informed consent compliant with ZIOPHARM policies and approved by the Human Investigation Review Committee with jurisdiction over the site;
4. ECOG performance score ≤ 1;
5. No chemotherapy, bortezomib, lenalidomide, thalidomide, arsenic trioxide, radiation therapy or immune therapy for ≥ 3 w and recovered from all treatment associated toxicities prior to registration; 5a. Patients may not receive more than the equivalent of 10 mg of prednisone per day for 2 weeks prior to registration.
6. Age ≥ 18;
7. Granulocytes ≥ 1.0 x 109/L; platelets ≥ 50 x 109/L;
8. Bilirubin ≤ 2.0 mg/dL; AST and ALT ≤ 2 x ULN;
9. Creatinine ≤ 3 X ULN.
10. No investigational agents within 28 days of study entry.
11. Males who agree to use a double-barrier method of birth control, (Double barrier method is defined as: a condom and either a diaphragm/cervical cap or an IUD).

Exclusion Criteria

1. NYHA functional class ≥ 3, myocardial infarction ≤ 6 mo or uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; QTc ≥ 450msec; AV-block ≥ grade-2 or LBBB;
2. Women of childbearing potential. (Non-childbearing potential is defined as: surgical sterilization or 2 years post-menopausal)
3. Active infection requiring antibiotics;
4. Allergy to ZIO-101 or its excipients;
5. Baseline confusion or dementia, defined as grade > 2 CTCAE Version 3.0;
6. Significant neurotoxicityneuropathology, defined as grade > 2 neurotoxicity neuropathology per CTCAE Version 3.0;
7. Prior seizures ≥ grade-3 in CTC v.3 criteria.
8. Prior history of neurological deficits (e.g., stroke, dementia, ischemia) that has the potential to confound a post-dose neurological assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 6 months

SECONDARY OUTCOMES:
Survival (overall and progression free) | 6 months
toxicities | 6 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Glendale, Arizona
  - Santa Barbara, California
  - Santa Rosa, California
  - West Hollywood, California
  - Bethesda, Maryland
  - Buffalo, New York
  - Charlotte, North Carolina
  - Sioux Falls, South Dakota